CLINICAL TRIAL: NCT03470077
Title: Effect of Intravenous Nalbuphine on Emergence Agitation in Children Undergoing Repair of Rupture Globe
Brief Title: Effect of Intravenous Nalbuphine on Emergence Agitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed abdelhameed, M.M.B.CH& Resident Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: postoperative EA in children
Record Dates: First submitted 2018-03-05; First posted 2018-03-19 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Nalbuphine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated into two groups of 40 patients each:
  Group A: will receive IV nalbuphine 0.1 mg/kg with induction of anesthesia. Group B: will receive IV nalbuphine 0.1 mg/kg at the end of surgery just before discontinuation of anesthesia.
Who Masked: Participant, Investigator
Masking Description: The trial will be planned that neither the doctors (investigators) nor the patients' guardians or even children themselves will be aware of the group allocation and timing of drug received
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 40 randomly allocated Patients undergoing repair of rupture globe will receive IV nalbuphine 0.1 mg/kg with induction of anesthesia.
  Interventions: Drug: IV nalbuphine 0.1 mg/kg with induction of anesthesia.
- Group B (Experimental): 40 randomly allocated Patients undergoing repair of rupture globe.will receive IV nalbuphine 0.1 mg/kg at the end of surgery just before discontinuation of anesthesia.
  Interventions: Drug: IV nalbuphine 0.1 mg/kg at the end of surgery.

INTERVENTIONS:
Drug: IV nalbuphine 0.1 mg/kg with induction of anesthesia. — Group A: 40 patients will receive IV nalbuphine 0.1 mg/kg with induction of anesthesia.
  .
  Other Names: nalufin
  Arms: Group A
Drug: IV nalbuphine 0.1 mg/kg at the end of surgery. — Group B: 40 patients will receive IV nalbuphine 0.1 mg/kg at the end of surgery just before discontinuation of anesthesia.
  Other Names: nalufin
  Arms: Group B

SUMMARY:
Our primary objective of this study is to compare the effect of administration of single dose of intravenous nalbuphine given with induction of anesthesia with intravenous nalbuphine given at the end of surgery on the incidence and severity of EA in children undergoing repair of rupture globe under general anesthesia.

The secondary outcomes will include FLACC score for postoperative pain assessment, hemodynamic variables, any complications as postoperative vomiting (POV) and sedation and parents' satisfaction score.

DETAILED DESCRIPTION:
Postoperative agitation, also referred to as emergence delirium is characterized by mental confusion, irritability, disorientation, inconsolable crying, and increased recovery time in the post anesthesia recovery room, increasing parents' concern and anxiety with respect to the clinical condition of their children . It can also lead to possible injury, damage to surgical dressings, lost intravenous catheters, disconnected cables and monitoring instruments, and source of dissatisfaction for parents, nurses, and others taking care of these children, and hence the children require extra nursing care and supplemental sedative and/or analgesic medications, which may delay patient discharge from hospital and are seven times more likely to have new-onset separation anxiety, apathy, and eating and sleep problems.

It is during the first 30 minutes after emergence that the greatest incidence of agitation is observed, and duration is generally limited and recovery occurs spontaneously. However, prolonged episodes of agitation lasting for up to 2 days have been described.

There is no definitive explanation for emergence agitation (EA). Many different causes have been suggested, such as rapid return of consciousness in an unfamiliar environment, the presence of pain (wounds, sore throat, and bladder distension), stressful induction, airway obstruction, a noisy environment, the duration of anesthesia, the child's personality, anesthetic premedication and the anesthetic technique used.

While its pathogenesis remains unclear, previous studies reported that ENT (ear, nose, and throat) surgical procedures have a higher incidence of EA in both adults and children . Children undergoing strabismus surgery under sevoﬂurane anesthesia often experience EA and postoperative vomiting (POV) .

Multiple medications including ketamine, propofol, clonidine, midazolam and fentanyl have been used effectively to prevent EA. However, these medications may increase sedation after anesthesia, cause slow awakening, and in some cases are associated with undesirable side effects, such as nausea and vomiting.

Nalbuphine is a synthetic opioid κ-receptor agonist μ-receptor antagonist with onset of action occurring within 2-3 min following IV injection, duration of analgesia of 3-6 hours and plasma half-life of 5 hours. Its analgesic potency approximately equals to morphine with less effects on cardiovascular and respiratory system, i.e., nalbuphine causes less intensive and less frequent decrease in blood pressure and respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-8 years.
* American Society of Anesthesiologists (ASA) physical status I-II scheduled to undergo repair of rupture globe.
* Gender: both.

Exclusion Criteria:

* Parent refusal.
* History of developmental delay or mental retardation.
* Known hypersensitivity to any drug used in this study.
* Children with co-morbid conditions like congenital heart disease, respiratory pathology and central nervous system disorders.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The incidence of Emergence Agitation in children undergoing repair of rupture globe under general anesthesia | at the first 30 minutes after surgery
  the Incidence of Emergence Agitation will be evaluated using Aono's four-point scale.
  * minimum score: 1
  * maximum score:4 Scores of one and two were considered as absence of EA, and scores of 3 and 4 were analyzed as presence of Emergence Agitation.
    1. Calm
    2. Not calm, but could be easily calmed
    3. Moderately agitated or restless
    4. Combative, excited, disoriente

SECONDARY OUTCOMES:
The severity of Emergency Agitation | at the first 30 minutes after surgery
  5- The severity of EA will be evaluated using the pediatric anesthesia emergence delirium scale A perfectly calm child scores 0 and extreme agitation corresponds to 20 points Agitation scores less than 10 will be interpreted as an absence of agitation, scores ≥ 10 will be regarded as presence of agitation, and scores ≥15 will be regarded as severe agitation
postoperative vomiting | first 48 hours after surgery
  Postoperative vomiting will be assessed using a numeric rank score
  * minimum score: 0
  * maximum score: 2 higher values represent a worse outcome and lowest values represent a better outcome 0 = no vomiting, 1 = vomited once, and 2 = vomited twice or more.
Postoperative sedation | first 48 hours after surgery
  Postoperative sedation will be assessed using sedation score described by Culebras et al (2001)
  * minimum score: 1
  * maximum score: 5 higher values represent a worse outcome and lowest values represent a better outcome 1. Awake and alert. 2. Sleeping but easily arouses to voice or light touch. 3. Arouses to loud voice or shaking. 4. Arouses with painful stimuli only. 5. Unarousable).
Postoperative FLACC Pain Score | first 24 hours after surgery
  Face, Legs, Activity, Cry, and Consolability (FLACC) pain score

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Abbas, Professor, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Vlajkovic GP, Sindjelic RP. Emergence delirium in children: many questions, few answers. Anesth Analg. 2007 Jan;104(1):84-91. doi: 10.1213/01.ane.0000250914.91881.a8. PMID 17179249
- [Background] Aono J, Ueda W, Mamiya K, Takimoto E, Manabe M. Greater incidence of delirium during recovery from sevoflurane anesthesia in preschool boys. Anesthesiology. 1997 Dec;87(6):1298-300. doi: 10.1097/00000542-199712000-00006. PMID 9416712
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Taddio A, Nulman I, Koren BS, Stevens B, Koren G. A revised measure of acute pain in infants. J Pain Symptom Manage. 1995 Aug;10(6):456-63. doi: 10.1016/0885-3924(95)00058-7. PMID 7561228
- [Background] Chen JY, Jia JE, Liu TJ, Qin MJ, Li WX. Comparison of the effects of dexmedetomidine, ketamine, and placebo on emergence agitation after strabismus surgery in children. Can J Anaesth. 2013 Apr;60(4):385-92. doi: 10.1007/s12630-013-9886-x. Epub 2013 Jan 24. PMID 23344921